CLINICAL TRIAL: NCT06158516
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial of Surufatinib as Adjuvant Therapy for Pancreatic Neuroendocrine Tumors
Brief Title: A Study of Surufatinib as Adjuvant Therapy for Pancreatic Neuroendocrine Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-NEN109
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — surufatinib

STUDY DESIGN:
Intervention Model Description: Arm A: surufatinib Arm B: placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib (Experimental)
  Interventions: Drug: Surufatinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300 mg once a day (QD) will be orally administrated on a 28-day cycle
  Arms: Surufatinib
Drug: Placebo — Placebo 300 mg once a day (QD) will be orally administrated on a 28-day cycle
  Arms: Placebo

SUMMARY:
pNENs still have a risk of recurrence after radical resection, and the overall recurrence and metastasis rate is as high as 13.7%-36.2% in China. At present, there is no standard adjuvant therapy for pNEN, and prospective studies are still lacking. This study was a randomized, double-blind, placebo-controlled, multicenter clinical trial to explore the efficacy and safety of surufatinib in the adjuvant treatment of pNET, in order to further improve the prognosis of patients and to provide high-quality research evidence for adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* pNETs lesions pathologically classified as WHO grade 1/ 2/ 3;
* G2/3-NET with at least one high-risk postoperative recurrence factor, including but not limited to lymph node metastasis, neurovascular invasion, pancreatic duct dilation, tumor >4cm, positive resection margin, etc.; or G1-NET with lymph node or remote transfer;
* Complete surgical resection (R0 or R1 was achieved) ;
* Adjuvant treatment was performed within 6-12 weeks after surgery;
* Have received whole-body 68Ga PET-CT examination within the past six months;

Exclusion Criteria:

* Urinalysis shows urine protein ≥ 2+ and 24-hour protein quantity test shows urinary protein ≥1 g;
* Under anti-hypertension treatment, still uncontrolled hypertension, defined as: systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg;
* Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina pectoris or coronary artery bypass grafting, congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular arrhythmias which needs drug treatment; LVEF (LVEF) <50%;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2026-11-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival (2y-DFS) | From the date of surgery to 2 years, assessed up to 24 months
  2-year disease-free survival (2y-DFS)

SECONDARY OUTCOMES:
Disease-free survival time | From the date of surgery to the date of distant metastasis or recurrence or death due to any cause, whichever came first, assessed up to 120 months
  Disease-free survival time
2-year Overall survival | From the date of surgery to 2 years, assessed up to 24 months
  2-year Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Doctor, Principal Investigator — Changhai Hospital; Jianming Xu, Doctor, Principal Investigator — Chinese PLA General Hosptial
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No